CLINICAL TRIAL: NCT05933993
Title: Mothers Experience of Pain Following Elective Cesarean Section. A Qualitative Study.
Status: Completed | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: Department of Regional Health Research, University of Southern Denmark, Odense, Denmark (Unknown); Department of Anesthesiology (4013), Copenhagen University Hospital, Copenhagen, Denmark (Unknown); Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Helene Korvenius Nedergaard, Primary investigator, Sygehus Lillebaelt
Other Study IDs: 979809337
Record Dates: First submitted 2023-06-21; First posted 2023-07-06 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section Complications
Keywords: postoperative pain; postoperative function; patient-relevant outcomes
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mothers, following an elective cesarean sections: The cohort in this study consists of Danish mothers, undergoing an elective cesarean section in one og the three participating hospitals.
  Interventions: Other: Elective cesarean section

INTERVENTIONS:
Other: Elective cesarean section — The study does not contain an intervention in itself, but women are included if they undergo an elective cesarean section

SUMMARY:
Background and aim:

In Denmark, approx 56.000 babies are born every year, and approx 20% of them are born by cesarean sections. Half of these cesarean sections are elective. Previous studies have shown that many women experience severe pain in the days following the cesarean section, thus limiting their ability to care for their baby and recover.

The Danish national anesthesiological research network, CEPRA (Collaboration for Evidence based Practice and Research in Anesthesia) is planning a national study on pain following elective cesarean sections. In order to assure that the investigators will be using actual patient-relevant outcomes in this large national study, the aim with this qualitative study is to obtain knowledge on how Danish women experience pain, recovery and function following an elective cesarean section.

Methods:

This is a qualitative study based on semi-structured telephone interviews with women 4-7 days after an elective cesarean section.

The study will take place in three Danish hospitals (Kolding, Copenhagen and Hillerød).

Women aged 18 or above, scheduled for elective cesarean section, will be eligible for inclusion.

Women will be informed about the study, orally and in writing, at the pre-anesthesiological consultation, which is held a few days before the cesarean section. Participation is completely voluntary. If they to participate, participants will sign a consent form. The investigators will include and interview participants until data saturation occurs. It is expected that 20-30 women should be included in total, evenly distributed at the three participating hospitals.

Interviews will be held by telephone, recorded digitally and transscribed verbatim. Transscribed interviews will be coded for categories and themes using the NVivo software. Data will be analysed using manifest content analysis.

Baseline characteristics will be handled with descriptive statistics.

The primary outcome of the study is a thematic analysis of Danish womens experience of pain, recovery and function following an elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing an elective cesarean section under spinal anesthesia
* speaking/writing Danish

Exclusion Criteria:

* cesarean section performed under general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Every person undergoing an elective cesarean section is eligible for inclusion.
Study Population: All adult women undergoing an elective cesarean section in one of the three participating hospitals are eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Pain | 4 to 7 days after the elective cesarean section
  The primary outcome of the study is a thematic analysis of Danish womens experience of pain following an elective cesarean section. As the study is qualitative, no scale will be used to measure pain, but instead the experience of pain as described by the participants.

SECONDARY OUTCOMES:
Recovery | 4 to 7 days after the elective cesarean section
  A secondary outcome of the study is a thematic analysis of Danish womens experience of recovery following an elective cesarean section. As the study is qualitative, no scale will be used, but instead the experience of recovery following cesarean section, as described by the participants
Physical function | 4 to 7 days after the elective cesarean section
  A secondary outcome of the study is a thematic analysis of Danish womens experience of physical function following an elective cesarean section. As the study is qualitative, no scale will be used, but instead the experience of physical function following cesarean section, as described by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Helene K Nedergaard, Principal Investigator — Lillebaelt Hospital Kolding, Department of Anesthesiology
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - North Zealand Hospital, Hillerød, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CEPRA, Collaboration for Evidence-based Practice and Research in Anesthesia — https://www.cepra.nu/